CLINICAL TRIAL: NCT02453451
Title: The Effect of the Iatrogenic Atrial Septal Defect After MitraClip Procedure on the Hemodynamic Outcome
Brief Title: The Effect of the Hole in the Cardiac Septum Developed by the MitraClip Procedure on the Blood Flow Mechanics
Acronym: MitraClipASD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 15-016
Record Dates: First submitted 2015-05-13; First posted 2015-05-25 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Atrial Septal Defect
Keywords: MitraClip; atrial septal defect; iatrogenic
MeSH Terms: conditions — Heart Septal Defects, Atrial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 2D-/3D-TTE; 3D-TEE, Walking Test (Experimental): 6 months after the MitraClip procedure
  Interventions: Other: 2D-/3D-TTE; Other: 3D-TEE; Other: Walking Test; Procedure: MitraClip procedure

INTERVENTIONS:
Other: 2D-/3D-TTE — recording of 3 cardiac cycles
  Other Names: 2-/3-dimensional transthoracic echocardiography
Other: 3D-TEE — with colour-Doppler techniques for recording the ASD and the mitral valve
  Other Names: 3-dimensional transesophageal echocardiogram
Other: Walking Test — for 6 minutes
Procedure: MitraClip procedure — catheter-based non-surgical procedure in which the atrioventricular valves were stuck together permanently via a clip (during the regular patient care)

SUMMARY:
Patients received a MitraClip procedure because of a leakiness of their mitral valves. During this procedure the atrioventricular valves were stuck together permanently via a clip which leads to a reduction of leakiness. As a result of this procedure a small hole remains at the cardiac septum which is called an atrial septal defect (ASD). In most cases the hole will close after a few weeks or months, but in many other cases not. Until now there is no exact data about the effect of this hole on the filling pressure in the heart or on the blood flow behaviour. So the aim of this study is a precise analysis of the blood flow mechanics during and after the MitraClip procedure to identify criteria to get more informations for a better strategy and regulation of the MitraClip procedure.

DETAILED DESCRIPTION:
The percutaneous mitral valve reconstruction (PMVR) using the MitraClip system has become an established therapeutic alternative for patients with symptomatic mitral regurgitation and high operative risk. The MitraClip technology represent a catheter-based non-surgical procedure in which a metal cramp (clip) is transported to the place of the defective mitral valve. At the same time, it occurs also a 3-dimensional transesophageal echocardiogram (3D-TEE) with a transseptal puncture to control this procedure. After removal of the guiding catheter a new atrial septal defect can develop which can close spontaneously after weeks or months.

In this study criteria for a standardized evaluation about the effect of the new ASD on hemodynamic parameters - before and after the MitraClip procedure - shall be validated for the first time. The investigators expect to obtain new findings through the exact analysis of the newly formed ASD for the planning, regulation and follow-up of the mitral insufficiency treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients in which a percutaneous mitral valve reconstruction via the MitraClip system shall be performed due to severe mitral insufficiency because a conventional surgery would be too stressful for them
* legal age (≥18 years)
* written informed consent prior to study participation
* subjects who are contractually capable and mentally able to understand and follow the instructions of the study personnel

Exclusion Criteria:

* malignant diseases
* varicose veins of the esophagus
* patients with central nervous system dysfunction
* pregnant and lactating females
* subject has been committed to an institution by legal or regulatory order
* dependency or working relationship with the investigator
* participation in a parallel interventional clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-07; Primary Completion 2017-01 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
change in hemodynamic parameters such as forward flow reduction through the mitral valve and left-to-right shunt due to the newly formed ASD | after 6 months

SECONDARY OUTCOMES:
quantitative change from baseline in the mitral regurgitation at 6 months | after 6 months
  2D and 3D transthoracic echocardiography (TTE) with colour-Doppler techniques
quality of life | after 6 months
  6 minutes walking test
change from baseline in the ASD area at 6 months | after 6 months
  3D TEE (Transesophageal echocardiogram) by direct en face imaging

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital RWTH Aachen, Department of Medical Clinic I, Aachen, Germany